CLINICAL TRIAL: NCT05916898
Title: Evaluation of the Safety and Efficiency of ShockWave Intravascular Lithotripsy (S-IVL) in Coronary Artery Diseases. The Lower Silesia Shockwave Registry (LSSR)
Brief Title: The Lower Silesia Shockwave Registry
Acronym: LSSR
Status: Recruiting | Type: Observational
Sponsor: Regional Cardiology Center, The Copper Health Centre (MCZ), (Other)
Collaborators: Provincial Specialized Hospital in Legnica (Unknown)
Responsible Party: Principal Investigator, Adrian Włodarczak, M.D.; Ph.D. Assoc Prof., Regional Cardiology Center, The Copper Health Centre (MCZ),
Other Study IDs: CopperHealthCentre
Record Dates: First submitted 2023-05-25; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Safety Issues; Efficacy, Self
Keywords: Percutaneous coronary interventions; Calcified Lesion; Shockwave intravascular lithotripsy; Stent under-expansion; Coronary artery diseases; lesion preparation; stent optimalization
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- S-IVL Intervention: Patients with the presence of a highly calcified, resistant lesion or a significantly under-expanded, previously implanted stent (regardless of the time of implantation) were part of the study cohort. The lesion was defined as resistant after an unsuccessful high-pressure NC balloon inflation (at least 20% under-expansion; whit at least 16 atm.). The decision regarding initial lesion preparation was left to the operators' dissertation and did not imply a recruitment process.
  There were no angiographic exclusion criteria regarding lesion anatomy regarding the length, tortuosity, severity, or prior stent placement. Operators supported by angiography assessment with optional intravascular imagining (IVUS/OCT) determined the size of the S-IVL catheter and an appropriate number of pulses for optimal vessel preparation or management of an under-expanded coronary stent.
  Interventions: Device: PCI with support of Shockwave Intravascular Lithotripsy

INTERVENTIONS:
Device: PCI with support of Shockwave Intravascular Lithotripsy — Coronary artery angioplasty of the primary lesion or optimization of the previously implanted stent with the support of Shockwave Intravascular Lithotripsy device

SUMMARY:
Lower Silesia Shockwave Registry (LSSR), is a observational registry collecting all consecutive cases of percutaneous coronary intervention (PCI) performed with the support of shockwave intravascular lithotripsy in two cooperating cardiac centers (Department of Cardiology, The Copper Health Centre, Lubin Poland, and Department of Cardiology, Provincial Specialized Hospital in Legnica, Poland).

DETAILED DESCRIPTION:
This study contains data from the Lower Silesia Shockwave Registry (LSSR), collecting all consecutive cases of percutaneous coronary interventions (PCI) performed with the support of shockwave intravascular lithotripsy from two cooperating cardiac centers (Department of Cardiology, The Copper Health Centre, Lubin Poland, and Department of Cardiology, Provincial Specialized Hospital in Legnica, Poland).

All patients involved in the study had a clinical indication for PCI based on current European Society of Cardiology (ESC) revascularisation guidelines, if necessary with the support of the local heart team.

Patients enrolled in the study had to meet one of two main inclusion criteria: The presence of a highly calcified, resistant lesion or a significantly under-expanded, previously implanted stent (regardless of the time of implantation). The lesion was defined as resistant after an unsuccessful high-pressure non-compliant (NC) balloon inflation (at least 20% under expansion; whit at least 16 atm.) The decision regarding initial lesion preparation was left to the operators' dissertation and did not imply a recruitment process. Patients meeting the inclusion criteria who initially underwent advanced debulking procedures (orbital or rotational atherectomy) were also recruited.

There were no angiographic exclusion criteria regarding lesion anatomy regarding the length, tortuosity, severity, or prior stent placement. Operators supported by angiography assessment with optional intravascular imagining (IVUS/OCT) determined the size of the S-IVL catheter and an appropriate number of pulses for optimal vessel preparation or management of an under-expanded coronary stent. Drug-eluting stent (DES) implantation or use of drug-eluting balloon catheters was left at the discretion of the operator.

The study had two primary endpoints- clinical success and safety outcome. The Clinical success was defined as an effective stent deployment or the optimization of previously not fully expanded stent (with less than <20% in-stent residual stenosis) [ and the presence of Thrombolysis in Myocardial Infarction (TIMI) 3 flow at the end of the procedure.

Safety outcomes were defined as procedural final serious angiographic complications procedural (perforation, abrupt closure, slow flow or no-reflow, unstable ventricular arrhythmias) and device failure (inability to cross the lesion, malfunction, or rapture). Also, adverse cardiac and cerebrovascular events (MACCE) were recorded. The MACCE consisted of death, myocardial infarction, acute cerebrovascular events, and repeated revascularization of the target lesion. Clinical follow-up was obtained by professional medical staff - personally or by telephone contacts periodically every 6 months after the index procedure. The study has the approval of a local ethics committee ( Bioethical Committee at the Lower Silesian Medical Chamber - number of approval 04/BOBD/2022).

ELIGIBILITY:
Inclusion Criteria:

* The presence of moderately to severely calcified lesions.
* The presence of significant under-expansion (greater than 20% of the diameter) of the previously implanted stent.
* Initial failure of the lesion preparation with either the NC balloon catheter or the atherectomy device.

Exclusion Criteria:

* Lack of patient consent
* Target vessel dissection type 3 or higher according to spontaneous coronary artery dissection (SCAD) classification
* Target vessel perforation due to previous unsuccessful lesion preparation
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-commers population with CAD treated by PCI performed with the support of shockwave intravascular lithotripsy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
The Clinical success | Evaluation at the end of index hospitalization
  Effective stent deployment or the optimization of previously not fully expanded stent (with less than <20% in-stent residual stenosis) and the presence of Thrombolysis in Myocardial Infarction (TIMI) 3 flow at the end of the procedure.
Incidence of Treatment-Emergent Adverse Events | Evaluation at the end of index hospitalization
  Safety outcomes were defined as procedural final serious angiographic complications procedural (perforation, abrupt closure, slow flow or no-reflow, unstable ventricular arrhythmias) and device failure (inability to cross the lesion, malfunction, or rapture).

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | Final assessment - 5 years after the initial hospitalization; followed by evaluation every 6 months from the end of the hospitalization until the final assessment (5 years).
  The MACCE consisted of death, myocardial infarction, acute cerebrovascular events, and repeated revascularization of the target lesion.

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Department of Cardiology, Provincial Specialized Hospital in Legnica,, Legnica, Lower Silesian Voivodeship
  - Department of Cardiology, The Copper Health Centre (MCZ), Lubin, Lower Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rola P, Wlodarczak A, Kulczycki JJ, Barycki M, Furtan L, Szudrowicz M, Jastrzebski A, Pecherzewski M, Doroszko A, Lesiak M. Feasibility of the intravascular lithotripsy in coronary artery disease. Short-term outcomes of the Lower-Silesia Shockwave Registry. Kardiol Pol. 2021;79(10):1133-1135. doi: 10.33963/KP.a2021.0093. Epub 2021 Aug 20. No abstract available. PMID 34415567